CLINICAL TRIAL: NCT05729269
Title: Characterization of Gut Microbiota in Chronic Liver Disease With Decreased Muscle Mass
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Dongtan Sacred Heart Hospital (Other); Hallym University Medical Center (Other); Hangang Sacred Heart Hospital (Other); Kangdong Sacred Heart Hospital (Other); Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: microbiota_CLD-sarcopenia
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2021-04

CONDITIONS: Gastrointestinal Microbiome; Sarcopenia; Liver Disease Chronic
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic liver disease: non-alcohol liver disease, alcohol liver disease, liver cirrhosis
  Interventions: Diagnostic Test: Sarcopenia_CT

INTERVENTIONS:
Diagnostic Test: Sarcopenia_CT — measurement of skeletal muscle through abdominal computed tomography

SUMMARY:
The purpose of this study was to confirm the presence of specific gut microbiota observed in patients with sarcopenia among patients who agreed to analyze gut microbiota through stool among multi-center chronic liver disease cohort patients.

DETAILED DESCRIPTION:
The effect of gut microbiota on liver disease is also well known and many studies are ongoing. A recently published study summarized the differences in the composition of gut microbiota in non-alcoholic fatty liver, steatohepatitis, and cirrhosis, and reported that metabolites from the changed gut microbiota may be a factor influencing non-alcoholic fatty liver disease (NAFLD) progression. These changes in gut microbiota composition have been reported to affect clinical outcomes in patients by causing an increase in endotoxin, a change in bile acid metabolism, and a decrease in short chain fatty acid. In particular, the reduction of short chain fatty acid is known to be associated with the occurrence of sarcopenia. Sarcopenia, which is common in patients with cirrhosis, which is a representative chronic liver disease, is well known as a poor prognostic factor for patients. Therefore, this study aims to analyze the distribution of gut microbiota observed in patients with sarcopenia through the gut microbiota investigated in the chronic liver disease cohort patient group and the characteristics of the distribution of gut microbiota for each disease corresponding to chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who have chronic liver disease (chronic liver disease cohort): alcohol liver disease, non-alcoholic liver disease, liver cirrhosis 2. Patients who consented to a study confirming the gut microbiota 3. Patients with abdominal computed tomography scan taken one month before or after submitting stool for gut microbiota analysis

Exclusion Criteria:

* Patients whose height and weight records are missing from the chart review

Ages: 24 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2017 to December 2019, 489 patients who agreed to collect feces among the cohort patients with chronic liver disease in five hospitals under the Hallym University Medical Center were surveyed.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fecal gut microbiota between sarcopenia group and non-sarcopenia group | 2 years
  Compare the species and proportions of the gut microbiota between sarcopenia group and non-sarcopenia group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Hallym University Medical College, Chuncheon, Gangwon-do, South Korea